CLINICAL TRIAL: NCT01827267
Title: A Phase 2 Study of Neratinib and Neratinib Plus Temsirolimus in Patients With Non-Small Cell Lung Cancer Carrying Known HER2 Activating Mutations
Brief Title: Neratinib With and Without Temsirolimus for Patients With HER2 Activating Mutations in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-NER-4201; 2012-004743-68 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-09 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: HER2-mutant Non-Small Cell Lung Cancer
Keywords: Lung cancer; Puma; neratinib; HKI-272; PB-272; Nerlynx
MeSH Terms: conditions — Lung Neoplasms | interventions — neratinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neratinib monotherapy (Experimental): 240 mg once daily with food, continuously in 21 day cycles
  Interventions: Drug: neratinib
- neratinib plus temsirolimus (Experimental): 240 mg neratinib plus 8 mg temsirolimus IV with optional dose escalation to 15 mg temsirolimus
  Interventions: Drug: neratinib; Drug: temsirolimus

INTERVENTIONS:
Drug: neratinib
  Other Names: Nerlynx
Drug: temsirolimus
  Other Names: Torisel
  Arms: neratinib plus temsirolimus

SUMMARY:
This is a Phase 2, therapeutic-exploratory, adaptive design, open-label, multicenter, multinational study evaluating neratinib monotherapy and neratinib plus temsirolimus combination therapy in patients with non-small cell lung cancer (NSCLC) who have documented somatic HER2 mutations.

DETAILED DESCRIPTION:
This is a Phase 2, therapeutic-exploratory, adaptive design, open-label, multicenter, multinational study evaluating neratinib monotherapy and neratinib plus temsirolimus combination therapy in patients with NSCLC and documented somatic HER2 mutations. Patients randomized at study entry into 1 of 2 treatment arms:

* Arm A: neratinib 240 mg orally once daily
* Arm B: neratinib 240 mg orally once daily plus temsirolimus 8 mg once weekly by intravenous (IV) infusion

In the case of disease progression, patients initially assigned to neratinib monotherapy arm given option to add temsirolimus 8 mg IV once weekly.

Patients on combination therapy given option to dose-escalate temsirolimus to 15 mg/week at the end of first cycle of treatment, if well tolerated and at the physician's discretion. If neratinib 240 mg/day plus temsirolimus 15 mg/week dose not well tolerated, patient subsequently dose reduced back to neratinib 240 mg/day plus temsirolimus 8 mg/week.

Dosing continuous on nominal 3-week cycles until evidence of progressive disease, unacceptable toxicity, or patient withdrawal of consent.

Disease measured radiographically at baseline and every 6 weeks until disease progression or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria

1. Aged ≥18 years at the time of signing the informed consent.
2. Histologically confirmed diagnosis of NSCLC, advanced (stage IIIB) or metastatic (stage IV).
3. Documented somatic ErbB2 (HER2) activating mutation.
4. Patients with anaplastic lymphoma kinase (ALK) translocations must have received crizotinib, except for cases of intolerable toxicity to crizotinib.
5. At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
6. Eastern Cooperative Oncology Group (ECOG) status <2.
7. Left ventricular ejection fraction (LVEF) ≥50% measured by multiple -gated acquisition scan (MUGA) or echocardiogram (ECHO).
8. Negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause.
9. Men and women of childbearing potential must agree and commit to the use of a highly effective method of contraception, as determined to be acceptable by the Investigator, from the time of informed consent until 3 months after the last dose of the investigational products.
10. Provide written, informed consent to participate in the study and follow the study procedures.

Exclusion Criteria

1. Previous treatment with any investigational agent ≤14 days prior to the initiation of investigational products.
2. Previous treatment with any strong inhibitor and/or inducer of CYP3A4 enzyme or sensitive P-glycoprotein (P-gp) substrates ≤30 days prior to the initiation of investigational products.
3. Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia.
4. Major surgery <30 days of starting treatment.
5. Chronic steroid use (prednisone >12.5 mg/day or dexamethasone >2 mg/day, excluding inhaled steroids).
6. Currently breast feeding.
7. Symptomatic or unstable brain metastases.
8. QTc interval >0.450 seconds for men and >0.470 seconds for women, or known history of QTc prolongation or Torsades de Pointes (TdP).
9. Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE v.4.0] diarrhea of any etiology at baseline).
10. Prior exposure to neratinib or mTOR inhibitor.
11. Active infection or unexplained fever >38.5°C (101.3°F).
12. Unable or unwilling to swallow tablets.
13. Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that would, in the Investigator's judgment, make the patient inappropriate for this study.
14. Known hypersensitivity to any component of the investigational products.
15. Unstable or uncontrolled diabetes mellitus (glycosylated hemoglobin [HbA1c] >6.5%).
16. Screening laboratory assessments outside the following limits: ANC <1000/μL (<1.0 x 109/L), Platelet count <75,000/μL (<75 x 109/L), Hemoglobin <8 g/dL, transfusions allowed, must be at least 7 days prior to baseline, Total bilirubin >1.5 x institutional upper limit of normal (ULN), AST and/or ALT 5 minutes, Creatinine clearance <50 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Senior Vice President, Study Director — Puma Biotechnology, Inc.
Locations (21):
- United States (15):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusettes General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- France (6):
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - CHRU de Lille - Hopital Calmette, Lille
  - Hopital Nord, Marseille
  - Hopitaux universitaires de Strasbourg Nouvel Hopital Civil, Strasbourg
  - CHU de Toulous Hopital Larre, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Li BT, Gandhi L, Ravichandran V, Besse B, Mazieres J, Shapiro GI, Boni V, Waqar SN, Park H, Quinn DI, Martinez A, Stemmer SM, Cortot AB, Barlesi F, Quoix E, Burkard ME, Selcuklu SD, Hunt C, Donoghue MTA, Kris MG, Bebchuk J, Eli LD, McCulloch L, Solit DB, Janne PA. Efficacy of Neratinib-Based Therapy in ERBB2-Mutant Lung Adenocarcinomas: Findings From 2 International Phase 2 Studies. Clin Lung Cancer. 2025 Oct 1:S1525-7304(25)00234-7. doi: 10.1016/j.cllc.2025.09.009. Online ahead of print. PMID 41193346

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib: Neratinib 240 mg
- Neratinib+Temsirolimus: Neratinib 240 mg + Temsirolimus 15 mg.
Period: Overall Study
Arm/Group | Neratinib | Neratinib+Temsirolimus
Started (Number of subjects randomized) | 18 (18 subjects were randomized but 17 received treatment.) | 44 (44 subjects were randomized; 43 subjects were treated.)
Received Study Drug | 17 | 43
Crossed Over to Neratinib + Temsirolimus | 11 | 0
Completed (Subjects completed study upon death.) | 13 | 32
Not Completed | 5 | 12
Not completed — Did not receive study drug | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Disease Progression | 1 | 1
Not completed — Sponsor Discontinued Study | 2 | 8
Not completed — Still on study | 0 | 2

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib | Neratinib+Temsirolimus | Total
Number analyzed (Participants) | 17 | 43 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 19 | 29
  >=65 years | 7 | 24 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.24 (8.88) | 63.44 (12.72) | 63.10 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 32 | 41
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as proportion of subjects who achieved confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  A complete or partial response must be confirmed no less than 4-weeks after the criteria for response are initially met.
Time Frame: From randomization to last tumor assessment, assessed up to 116.5 weeks. For the Neratinib arm, only tumor assessments prior to crossover were included.
Population: All subjects who received at least 1 dose of drug
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib | Neratinib+Temsirolimus
Number analyzed (Participants) | 17 | 43
Participants | 0 | 6

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the proportion of patients who achieved objective response (CR or PR) or stable disease (SD) for at least 12 weeks.
Time Frame: as for outcome 1
Population: All subjects who received at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib | Neratinib+Temsirolimus
Number analyzed (Participants) | 17 | 43
Participants | 6 | 21

3. Secondary Outcome: Duration of Response (DOR)
Description: Measured from the time at which measurement criteria were first met for CR or PR (whichever status was recorded first), until the date of first recurrence, progressive disease (PD), or death was objectively documented, taking as a reference for PD the smallest measurements recorded since enrollment, per RECIST (v1.1) criteria.
Time Frame: as for outcome 1
Population: All subjects who received at least 1 dose of drug and had either complete or partial response.
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib | Neratinib+Temsirolimus
Number analyzed (Participants) | 0 | 6
Participants
  Less than 3 months | 0 | 2
  3 to less than 6 months | 0 | 2
  6 to less than 12 months | 0 | 0
  Greater than 12 months | 0 | 2

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as time from date of randomization until the first disease recurrence or progression per RECIST V1.1 or death due to any cause; censored at the last assessable evaluation or at the initiation of new anti-cancer therapy. Disease assessment is based on investigator tumor assessments. If no post-baseline tumor assessment then censored at enrollment date.
Time Frame: as for outcome 1
Population: All subjects who received at least 1 dose of drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Neratinib+Temsirolimus
Number analyzed (Participants) | 17 | 43
months | 2.9 [1.4 to 9.8] | 4.0 [2.9 to 5.4]

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time (month) from randomization to death due to any cause; censored at the date last known alive.
Time Frame: From randomization to death or end of long term follow-up, assessed up to 31.8 months.
Population: All subjects who received at least 1 dose of drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neratinib | Neratinib+Temsirolimus
Number analyzed (Participants) | 17 | 43
months | 10.0 [4.9 to 18.9] | 15.1 [10.8 to 17.7]

ADVERSE EVENTS:
Time Frame: From time of first dose through 28 days after last dose, assessed up to 116.5 weeks.
Groups:
- Ner+Tem Post Crossover: Neratinib 240 mg + Temsirolimus 15 mg for subjects who crossed over from Neratinb 240 mg arm
Arm/Group | Neratinib | Neratinib+Temsirolimus | Ner+Tem Post Crossover
Serious Adverse Events (participants affected / at risk) | 7/17 | 16/43 | 7/11
Other Adverse Events (participants affected / at risk) | 17/17 | 43/43 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=17) | Neratinib+Temsirolimus (N=43) | Ner+Tem Post Crossover (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Pachymeningitis (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=17) | Neratinib+Temsirolimus (N=43) | Ner+Tem Post Crossover (N=11)
Anaemia (Blood and lymphatic system disorders) | 5 | 18 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1
Vision blurred (Eye disorders) | 0 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 8 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Cheilosis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 18 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 37 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 4 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 24 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 21 | 2
Vomiting (Gastrointestinal disorders) | 5 | 14 | 1
Asthenia (General disorders) | 6 | 12 | 1
Catheter site erythema (General disorders) | 1 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 2 | 0
Chills (General disorders) | 3 | 5 | 1
Fatigue (General disorders) | 4 | 17 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 1
Nodule (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 7 | 0
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 2
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 1
Rhinitis (Infections and infestations) | 0 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 4 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 10 | 0
Amylase increased (Investigations) | 2 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 10 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 1
Blood creatinine increased (Investigations) | 1 | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 3 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 5 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 10 | 1
White blood cell count decreased (Investigations) | 1 | 5 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 23 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 7 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 13 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 8 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 13 | 1
Headache (Nervous system disorders) | 2 | 10 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 2
Insomnia (Psychiatric disorders) | 1 | 7 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 6 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 4 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 10 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 12 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less